CLINICAL TRIAL: NCT01407809
Title: Venous Sinus Stenting for Idiopathic Intracranial Hypertension Refractory to Medical Therapy
Acronym: VSSIIH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1004011008
Record Dates: First submitted 2011-06-13; First posted 2011-08-02 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Idiopathic Intracranial Hypertension (IIH)
MeSH Terms: conditions — Pseudotumor Cerebri

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Intervention (Experimental)
  Interventions: Device: Venous Sinus Stenting

INTERVENTIONS:
Device: Venous Sinus Stenting — Venous sinus stenting consists of placing a stent into the narrowed veins of the brain.

SUMMARY:
Idiopathic Intracranial Hypertension (IIH) is a disease that affects mainly young people, and is associated with headache and loss of vision. The medical and surgical management of IIH is problematic and many patients are not treated effectively. Some cases of IIH are associated with severe stenosis of the large veins of the brain and various researchers have recently reported significant improvement in patients with IIH after the narrow veins of the brain were treated with a stent. Our project aims to evaluate the safety and long-term efficacy of venous sinus stenting in patients with severe IIH refractory to medical management.

ELIGIBILITY:
INCLUSION CRITERIA

1. Age > 18 years
2. Established diagnosis of Idiopathic Intracranial Hypertension according to the criteria of the 2004 International Classification of Headache Disorders (Table 3).
3. Visual field loss: One of criteria A, B or C must be fulfilled.

   A. Severe visual function loss, defined as grades 4 and 5 on the Humphrey Visual Field Analyzer SITA Standard 24-2 Test grading scale (Table 4) at initial presentation.

   B. Moderate visual function loss, defined as grade 3 on the Humphrey Visual Field Analyzer SITA Standard 24-2 Test grading scale (Table 4) at presentation and failure of treatment with acetazolamide (Diamox) given at efficient dose (2g/d or maximum tolerated dose) or Topiramate (Topamax) given at efficient dose (maximum 150mg daily). Failure is defined by the absence of visual function improvement after 1 month of treatment and/or medication intolerance.

   C. Mild visual function loss, defined as grades 0,1 or 2 on the Humphrey Visual Field Analyzer SITA Standard 24-2 Test grading scale (Table 4) at presentation and a worsening to moderate or greater visual function loss, defined as grades 3-5, after 1 month of treatment and/or medication intolerance.
4. Magnetic Resonance Venography (MRV) or Computed Tomography Venography (CTV) demonstrating bilateral transverse sinus stenosis or unilateral transverse sinus stenosis with contralateral transverse sinus hypoplasia or atresia. At least one of the stenoses must cause ≥ 50% reduction of the sinus lumen diameter.
5. Signed informed consent obtained from the patient.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-01; Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Absence of procedure related and device related complications. | 24 months
Clinically significant cerebrospinal fluid (CSF) pressure reduction AND improvement of more than one grade in the Humphrey Field SITA Standard 24-2 Test grading scale. | 24 months
Greater than 2 decibel (dB) mean deviation compared to the pre-operative field testing. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Athos Patsalides, MD, MPH, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- New York Presbyterian/ Weill Cornell Medicine, New York, New York, United States

REFERENCES:
- [Derived] Boddu SR, Gobin YP, Dinkin M, Oliveira C, Patsalides A. Impaired drainage of vein of Labbe following venous sinus stenting for idiopathic intracranial hypertension. J Neurointerv Surg. 2019 Mar;11(3):300-306. doi: 10.1136/neurintsurg-2018-014153. Epub 2018 Sep 15. PMID 30219791